CLINICAL TRIAL: NCT02079558
Title: Efficacy of Oxytocin vs. Carbetocin in Prevention of Postpartum Hemorrhage After Cesarean Section
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Dr Robabeh Taheripanah, Associated prof. Obstetrics & Gynecology, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: IRHRC-021; JANU2014TAHERIPANAH
Record Dates: First submitted 2014-01-13; First posted 2014-03-06 (Estimated); Last update posted 2014-03-06 (Estimated); Status verified 2014-03

CONDITIONS: Postpartum Hemorrhage
Keywords: prevention; cesarean section
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — carbetocin; Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxytocin (Experimental): A single 100 microgram IV dose of carbetocin after operation
  Interventions: Drug: Oxytocin
- Carbetocin (Experimental): A standard 30 international units (IU) IV infusion of oxytocin during two hours
  Interventions: Drug: Carbetocin

INTERVENTIONS:
Drug: Carbetocin — Carbetocin with single 100 microg IV dosage was used in this investigation
  Other Names: Duratocin,; Pabal,; Lonactene
  Arms: Carbetocin
Drug: Oxytocin — Oxytocin with 30 international units (IU) IV infusion was used in this investigation
  Other Names: Pitocin
  Arms: Oxytocin

SUMMARY:
Postpartum hemorrhage (PPH) is a common complication of childbirth and a leading cause of maternal morbidity and mortality. The prompt and effective treatment of subjects with PPH would reduce operation risks. Hence in this study, the efficacy of Oxytocin and Carbetocin was compared in prevention of postpartum hemorrhage after cesarean sections.

ELIGIBILITY:
Inclusion Criteria:

* At least one risk for postpartum hemorrhage and lack of hypersensitivity to oxytocin and carbetocin

Exclusion Criteria:

* Patients' refusal to cooperate, major therapeutic side effects, history of cardiac and renal disease or preeclampsia

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
screening of Cessation of bleeding | screening until 24 hours after placenta disconnection
time duration to stop bleeding in the case of post-cesarean section | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Robabeh Taheripanah, MD-Gyn., Principal Investigator — Infertility and Reproductive health Research center, Imam Hossien hospital, Shahid Beheshti Medical university, Tehran, Iran
Locations (1):
- Infertility and Reproductive Health Research Center, Tehran, Tehran Province, Iran

REFERENCES:
- [Derived] Taheripanah R, Shoman A, Karimzadeh MA, Zamaniyan M, Malih N. Efficacy of oxytocin versus carbetocin in prevention of postpartum hemorrhage after cesarean section under general anesthesia: a prospective randomized clinical trial. J Matern Fetal Neonatal Med. 2018 Nov;31(21):2807-2812. doi: 10.1080/14767058.2017.1355907. Epub 2017 Jul 25. PMID 28707488